CLINICAL TRIAL: NCT05828979
Title: Feasibility sTudy to Assess the URoMems Artificial uriNary Sphincter In the Treatment of Stress Incontinence in wOmeN
Brief Title: Clinical Investigation to Assess a New Artificial Urinary Sphincter to Treat Urinary Incontinence in Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UroMems SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP CCH2211240956
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Urinary Incontinence,Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- UroMems artificial urinary sphincter (Experimental): Female adults (18+) with urinary incontinence with reduced outlet resistance due to intrinsic sphincter deficiency.
  Interventions: Device: UroMems artificial urinary sphincter

INTERVENTIONS:
Device: UroMems artificial urinary sphincter — Implantation of the device

SUMMARY:
Prospective multicenter study designed to test the feasibility of the UroMems Artificial Urinary Sphincter in women

DETAILED DESCRIPTION:
This study is a prospective, open-label, non-randomized, multi-center, single-arm, study with subjects acting as their own control designed to test the feasibility of a new artificial urinary sphincter the UroMems eAUS (investigational name of device called UroActive) in women.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years old
* Female patient
* Cognitively able and willing to sign an informed consent
* Stable medication regimen (including prescription, over the counter, and supplements) for the past 3 months
* Use of medically acceptable contraception, if of childbearing potential
* Able and willing to comply with follow-up investigations, including maintaining consistent medication use and fluid intake through the primary endpoints
* Has adequate cognitive and manual capabilities to operate the UroMems eAUS System as assessed by the investigator
* Is an appropriate surgical candidate and has no medical or mental condition that would interfere with study procedures or confound study outcomes as assessed by the investigator
* Life expectancy ≥ 5 years as assessed by the investigator
* Affiliated with an appropriate social security system
* Has failed or is not a candidate for other treatments for urinary incontinence, either surgical or conservative, including slings, ACT, etc. (excluding other AUS devices)
* Negative urine culture prior to the procedure
* Urinary incontinence assessed by investigator with at least ≥ 50 g in 24-hour pad-weight tests
* Clinically insignificant post-void residual (PVR) urine defined as < 50 ml and/or no greater than 10% of the voided volume
* Complains of urine leakage on coughing, laughing, and/or moving and/or presence of orthostatic urine leakage by self-report as recorded in baseline bladder diary

Exclusion Criteria:

* Currently enrolled or plans to enroll in another investigational device or clinical drug trial or has completed an investigational study within 3 months
* Vulnerable patient (patient deprived of their liberty due to a judicial or administrative decision, patient suffering from psychiatry troubles preventing her from giving her consent, patients hospitalized for reason other than the current clinical investigation, patient under 18 years of age, patient under tutelage, patient having withdrawn her consent)
* Patients whom the investigator determines to be poor candidate for surgical procedures and/or anesthesia due to physical or mental conditions
* Pregnant patient, or patient planning pregnancy during the study duration
* Patient presenting one or several contraindications of the device
* Any planned procedure requiring urethral catheterization 12 months after implant procedure (include intermittent catheterization) except for diagnostic purposes
* Known allergy to UroMems eAUS implantable components
* History of pelvic irradiation (external beam therapy or brachytherapy)
* Uncontrolled diabetes mellitus defined as persistent blood sugar level recordings of >12 mmol/l (216 mg/dl) and a glycosylated hemoglobin (HbA1C) of >9% (75 mmol/mol) over the preceding 3 months
* History of bleeding diathesis or cannot stop usage of an anti-coagulant until the International Normalized Ratio (INR) is below 1.5 or quick value >70
* Any genito-urinary malignancies which are not in remission for at least 2 years or considered cured
* Previous AUS implant
* Currently has another Active Implantable Medical Device (AIMD) implanted
* Urge incontinence, mixed incontinence (MI) with a predominant urgency component
* Overflow urinary incontinence
* Neurogenic bladder dysfunction that is not treatable or controllable by pharmacological or any alternative methods
* Abnormal or poor bladder compliance defined as being <30 ml/ cm H2O
* Bladder neck or urethral stricture that may require any long-term instrumental treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Rate of explants and revisions at 6 months after device activation | 6 months after device activation
  Rate of explants and revisions
Rate of device activation successes | 5 weeks after device implantation
  Rate of device activation successes

SECONDARY OUTCOMES:
Number of subjects with 50% reduction or greater in 24-hour pad weight test | 90, 185 and 365 days after activation
  Number of subjects with 50% reduction or greater in 24-hour pad weight test
Number of subjects with 75% reduction or greater in 24-hour pad weight test | 90, 185 and 365 days after activation
  Number of subjects with 75% reduction or greater in 24-hour pad weight test
3-day bladder diary | 90, 185 and 365 days after activation
  Bladder diary will be filled in during 3 consecutive days
General quality of life questionnaire | 90, 185 and 365 days after activation
  General quality of life questionnaire
Disease specific questionnaire (level of incontinence) | 90, 185 and 365 days after activation
  Disease specific questionnaire (level of incontinence)
Disease specific questionnaire (symptoms and quality of life) | 90, 185 and 365 days after activation
  Disease specific questionnaire (symptoms and quality of life)
Disease specific questionnaire (sexual activity) | 90, 185 and 365 days after activation
  Disease specific questionnaire (sexual activity)
Disease specific questionnaire (quality of life) | 90, 185 and 365 days after activation
  Disease specific questionnaire (quality of life)
Disease specific questionnaire (type of incontinence) | 90, 185 and 365 days after activation
  Disease specific questionnaire (type of incontinence)
Post void residuals | Baseline, within 45 days after baseline (device implantation), 14 days after implantation, 5 weeks after implantation (device activation), and 14, 30, 90, 185, 365 and 730 days after activation
  Post void residuals will be measured to assess the bladder function
Patient satisfaction | 5 weeks after device implantation (device activation), and 14, 30, 90, 185, 365 and 730 days after activation
  Patient satisfaction questionnaire
Physician satisfaction questionnaire | Within 45 days after baseline (device implantation), 5 weeks after implantation (device activation), and 14, 30, 90, 185, 365 and 730 days after activation
  Questionnaire to assess the physician satisfaction regarding the procedure and the device
Rate of adverse events | Baseline, within 45 days after baseline (device implantation), 14 days after implantation, 5 weeks after implantation (device activation), and 14, 30, 90, 185, 365 and 730 days after activation
  All categories: serious/not serious events and device- and procedure-related effects

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Chartier-Kastler, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière
Locations (2):
- France (2):
  - CHU Nantes, Nantes
  - Groupe Hospitalier Pitié-Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: No